CLINICAL TRIAL: NCT03646110
Title: The Comparison of Single and Multi-incision Minimally Invasive Esophagectomy for Treating Esophageal Cancer
Brief Title: The Comparison of Single and Multi-incision MIE for Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201804074RINA
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; Minimally invasive esophagectomy (MIE); single-incision Minimally invasive esophagectomy (SIMIE)
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-incision MIE (Experimental): Esophageal cancer patients received single-incision Minimally invasive esophagectomy
  Interventions: Procedure: Minimally invasive esophagectomy
- multi-incision MIE (Active Comparator): Esophageal cancer patients received multi-incision Minimally invasive esophagectomy
  Interventions: Procedure: Minimally invasive esophagectomy

INTERVENTIONS:
Procedure: Minimally invasive esophagectomy — Minimally invasive esophagectomy is a surgical procedure for esophageal resection

SUMMARY:
Minimally invasive esophagectomy (MIE) has been gradually adopted as a feasible and effective treatment option for esophageal cancer. Previously the investigators have published the adoption of single-incision approach both in the thoracoscopic and laparoscopic phases in MIE (SIMIE).The preliminary clinical results showed that SIMIE can provide an equivalent perioperative outcome whereas reduced the wound pain on the days 7 after surgery as compared to MIE performed with multi-incision (MIMIE). The goal of the current study was to conduct a prospective randomized trial to compare the perioperative outcome and survival of SIMIE and MIMIE.

DETAILED DESCRIPTION:
Surgery remains the main stay of treating esophageal cancer. However, esophagectomy is a complex and technical demanding surgical procedure harboring substantial morbidity and mortality. Minimally invasive esophagectomy (MIE) has been gradually adopted as a feasible and effective treatment option for esophageal cancer. The standardized procedure including lymph node dissection, esophageal mobilization and reconstruction can be effectively performed under minimized wound incision whereas rendering the patients a possibility of faster postoperative recovery and reduced risk of perioperative postoperative pulmonary complication. The procedure of MIE including the thoracoscopic and laparoscopic phases which are usually performed multiple incisional wounds. Previously the investigators have published the adoption of single-incision approach both in the thoracoscopic and laparoscopic phases in MIE (SIMIE). The preliminary clinical results showed that SIMIE can provide an equivalent perioperative outcome whereas reduced the wound pain on the days 7 after surgery as compared to MIE performed with multi-incision (MIMIE). The goal of the current study was to conduct a prospective randomized trial to compare the perioperative outcome and survival of SIMIE and MIMIE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of esophageal cancer
2. Age between 35 to 75 years old
3. Resectable tumor as evaluation by preoperative imaging studies.

Exclusion Criteria:

1. Previous surgery in the chest or abdomen.
2. Receiving definitive chemoradiation (5500 cGy or more).
3. Tumor invasion to the trachea, spine or aorta.
4. Liver cirrhosis with esophageal varices or liver cirrhosis refractory to medical treatment, Child C classification.
5. Previous history of cerebral vascular attack.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2021-07-26 (Estimated); Study Completion 2021-07-26 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 60 months
  Overall survival rate of the participants after surgery

SECONDARY OUTCOMES:
Pain score as assessed by the face rating scale | 1,7,14,28 days
  The scale range of face rating scale is ranging from 0 (happy face) to 10 (crying face). Higher values represent a worse outcome.
Ratio of ambulation | post-operative day 2 (POD2)
  30-minute walk test
Postoperative force vital capacity | 1 and 3 months
  Force vital capacity (FVC) is one of the most common parameters for pulmonary function measured in spirometry
Post operative forced expiratory volume in one second | 1 and 3 months
  Forced expiratory volume in one second (FEV1) is one of the most common parameters for pulmonary function measured in spirometry
Postoperative pulmonary complication | 1 month
  pulmonary complication after esophagectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Jang-Ming Lee, Taipei, Zhongzheng Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: previous SIMIE study 1 — http://www.ncbi.nlm.nih.gov/pubmed/26547093
- See also: previous SIMIE study 2 — http://www.ncbi.nlm.nih.gov/pubmed/27826778